CLINICAL TRIAL: NCT06460129
Title: Effects of Bruegger's Versus Kendall Exercises on Pain, Range of Motion, Craniovertebral Angle and Functional Disability in Patients With Cervical Postural Syndrome
Brief Title: Effects of Bruegger's Versus Kendall Exercises in Cervical Postural Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/23/01105
Record Dates: First submitted 2024-06-11; First posted 2024-06-14 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Neck Pain
Keywords: Bruegger's exercises; Kendal exercises; Forward Neck Posture; Mobile Posture
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Brugger's Exercises (Experimental): Participants will receive Burger Exercise
  Interventions: Other: Brugger's Exercises
- KENDALL EXERCISE (Active Comparator): Participants will receive Kendal Exercise
  Interventions: Other: Kendal Exercise

INTERVENTIONS:
Other: Brugger's Exercises — 1. The participant will sit upright and wrap an elastic resistance band around each hand, leaving the palms open. They will perform thumb and finger abduction and extension, wrist extension, and forearm supination. This will be followed by scapular retraction with shoulder external rotation, elbow extension, shoulder abduction, and extension, holding this position for 10 seconds.
  2. In both sitting and standing positions, the participant will sit at the edge of a seat, naturally lifting the sternum, with legs spread at a 45-degree angle and feet slightly turned out. Shoulders should be relaxed, chin tucked, and elbows fully extended. The participant will keep their shoulders down, imagining the scapulae pressing together and downward into a V shape, with thumbs turned out, palms up, and fingers spread. This position is held for 10 seconds.
  Arms: Brugger's Exercises
Other: Kendal Exercise — 1. In a supine position, the participant will place a towel around their neck. With their head on the floor, they will tuck their chin and use the towel to apply gentle resistance, holding for 10 seconds to strengthen the deep flexor muscles of the cervical spine.
  2. In a prone position, the participant will point their thumbs toward the ceiling and extend their arms fully while leaning forward, then return to the starting position. They will then extend their arms horizontally and hold for 10 seconds.
  3. The participant will place both hands on the back of their head, lift their elbows upward, pull them back, and simultaneously spread their arms out to the side. This position will be held for 10 seconds before returning to the starting position.
  Arms: KENDALL EXERCISE

SUMMARY:
Cervical Postural Syndrome is an uncomfortable and painful condition characterized by a protruding chin and rounded shoulders, commonly resulting from poor posture in the neck, middle back, and shoulders. This syndrome often leads to an excessive forward curvature of the upper back, causing the chin to jut forward and the shoulders to hunch forward. A prevalent cervical abnormality associated with this condition is the forward head position, which increases the risk of neck pain. The entire clinical condition is referred to as "sterno-symphyseal syndrome" by Bruegger. He describes the muscles involved as "painfully tense and painfully weak." Bruegger's exercises are designed to align the spine correctly by strengthening the scapular and neck muscles. Similarly, Kendall's exercises focus on restoring cervical spine alignment, particularly for individuals with forward head posture, by targeting the shoulder extensors and deep neck flexors. While numerous studies have examined the direct effects of forward head posture on the cervical spine, there is limited research comparing the effectiveness of Bruegger's exercises and Kendall's exercises, particularly regarding exercises that do not directly target the neck.

DETAILED DESCRIPTION:
Cervical Postural Syndrome is a common and painful condition characterized by a projecting chin and rounded shoulders, resulting from poor posture in the neck, middle back, and shoulders. This syndrome often causes an exaggerated forward curvature of the upper back, leading to a forward-protruding chin and forward-sitting shoulders. The forward head position is a prevalent cervical issue that increases the risk of neck pain. Bruegger refers to this condition as "sterno-symphyseal syndrome," describing the involved muscles as "painfully tense and painfully weak." Bruegger's exercises aim to correct spinal alignment by strengthening the scapular and neck muscles. Kendall's exercises focus on restoring cervical spine alignment, especially for those with forward head posture, by strengthening the shoulder extensors and deep neck flexors. While many studies have examined the direct impact of forward head posture on the cervical spine, there is limited research comparing the effectiveness of Bruegger's exercises and Kendall's exercises, particularly for exercises that do not directly target the neck.

The objective of this study will be to compare the effects of Bruegger's exercises and Kendall's exercises on pain, range of motion, craniovertebral angle, and functional disability in patients with Cervical Postural Syndrome.

A randomized clinical trial will be conducted at Rasheed Hospital, using a non-probability convenient sampling technique on 36 patients who will be divided into two groups. One group will follow the Bruegger's exercises protocol, while the other group will follow Kendall's exercises. The protocol duration will be six weeks, with sessions three times a week. Each session will consist of one set of 10 repetitions for each movement, repeated for three sets, with a 10-second rest per repetition, a one-minute rest after each set, and a three-minute rest between each movement. Outcome measures will include pain, range of motion, craniovertebral angle, and functional disability. Data will be collected before and after the training sessions. The data will be entered and analyzed using SPSS version 25, and the Shapiro-Wilk test will be applied to determine the normality of the data.

ELIGIBILITY:
Inclusion Criteria:

* Age range: 20-40
* A patient who has neither "specific pain" nor "poor posture."
* A cranio-vertebral angle (CVA) of less than 52 degrees
* A Numeric Pain Rating Scale (NPRS) score of fewer than 7
* A Neck Disability Index score of greater than 10 (NDI)

Exclusion Criteria:

* Surgery on the neck or back
* Recent trauma history
* Malignancy
* Cervical dysfunction-related neurological symptoms
* Temporomandibular joint surgery
* Recent fractures or injuries

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2024-12-15 (Actual); Primary Completion 2025-04-15 (Actual); Study Completion 2025-05-07 (Actual)

PRIMARY OUTCOMES:
Pain level | 6th week
  A numerical pain rating scale is a quantitative tool for determining how much pain is experienced. This scale is trustworthy and valid for measuring pain. Its measurement ranges from 0 to 10. I mean that when the numbers go from 0 to 10, the pain is more intense. O denotes "no pain," 1-3 indicate "mild pain," 4-6 indicate "moderate pain," 7-9 indicate "severe pain," and 10 indicate the worst pain. Dependability
Range of Motion | 6th week
  Range of movement refers to the area that a joint can cover while moving. We utilize a universal goniometer to measure the range of motion (ROM). A scale called a universal goniometer is used to measure the range of quantitative values. The universal goniometer is also a useful and trustworthy instrument for ROM measurement. For cervical range of motion and cranio-vertebral angle, therefore, we use it.
limited function | 6th week
  Disability is the inability of an individual to accomplish a goal or to carry out a daily activity. The Neck Disability Index (NDI) is the main tool used in neck assessments. The NDI is a scale used to assess a joint's limited range of motion or to measure the
  useful action. This scale has ten items that are linked to carrying out an activity. The neck impairment can be measured using this accurate and trustworthy scale. Dependability

CONTACTS AND LOCATIONS:
Overall Officials: Arslan Qaramat, DPT, Principal Investigator — Riphah International University
Locations (1):
- Rasheed Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Avaghade RR, Shinde SB, Dhane SB. Effectiveness of McKenzie approach and segmental spinal stabilization exercises on neck pain in individuals with cervical postural syndrome: An experimental study. J Educ Health Promot. 2023 Jul 29;12:225. doi: 10.4103/jehp.jehp_239_23. eCollection 2023. PMID 37727425
- [Background] Abdel-Aziem AA, Abdel-Ghafar MA, Ali OI, Abdelraouf OR. Effects of smartphone screen viewing duration and body position on head and neck posture in elementary school children. J Back Musculoskelet Rehabil. 2022;35(1):185-193. doi: 10.3233/BMR-200334. PMID 34092602
- [Background] Kazeminasab S, Nejadghaderi SA, Amiri P, Pourfathi H, Araj-Khodaei M, Sullman MJM, Kolahi AA, Safiri S. Neck pain: global epidemiology, trends and risk factors. BMC Musculoskelet Disord. 2022 Jan 3;23(1):26. doi: 10.1186/s12891-021-04957-4. PMID 34980079
- [Background] Al-Khazali HM, Younis S, Al-Sayegh Z, Ashina S, Ashina M, Schytz HW. Prevalence of neck pain in migraine: A systematic review and meta-analysis. Cephalalgia. 2022 Jun;42(7):663-673. doi: 10.1177/03331024211068073. Epub 2022 Feb 15. PMID 35166137
- [Background] Richards KV, Beales DJ, Smith AL, O'Sullivan PB, Straker LM. Is Neck Posture Subgroup in Late Adolescence a Risk Factor for Persistent Neck Pain in Young Adults? A Prospective Study. Phys Ther. 2021 Mar 3;101(3):pzab007. doi: 10.1093/ptj/pzab007. PMID 33444448